CLINICAL TRIAL: NCT01017445
Title: Boonme Stick Exercise vs. Quadriceps Strengthening Exercise in Knee Osteoarthritis : A Randomized Controlled Trial
Brief Title: Stick Versus Quadricep Exercise for Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Boonsin Tangtrakulwanich, Department of Orthopaedic surgery, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 50/369-011
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis, exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quadricep strengthening exercise (Experimental): Quadricep strengthening exercise
  Interventions: Other: Boonme stick exercise

INTERVENTIONS:
Other: Boonme stick exercise — individual exercise daily

SUMMARY:
This study aims to compare the efficacy between Boonme stick exercise and quadriceps strengthening exercise in knee osteoarthritis.Patients diagnosed as knee osteoarthritis using Altman criteria will be randomized into 2 groups using simple random technique. Patients will be instructed and trained for both quadriceps or Boonme stick exercise by one-trained physical therapist. All patients will be treated with behavioral modification, NSAIDs and analgesic drugs and regularly follow-up . Assessment included visual analogue scale, exercise compliance, WOMAC and patient satisfaction were done by an assessor in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis using Altman criteria

Exclusion Criteria:

* problem of communication ability

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
vas score | 1,2 years

SECONDARY OUTCOMES:
WOMAC | 1,2 yrs
number of analgesic used | 1,2 years

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD.,Ph.D, Principal Investigator — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand